CLINICAL TRIAL: NCT05500170
Title: The Benefits of Nicotinamide Riboside Upon Cognition and Sleep in Older Veterans
Brief Title: Benefits of Nicotinamide Riboside Upon Cognition and Sleep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Carleara Weiss, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FP00006694
Record Dates: First submitted 2022-08-09; First posted 2022-08-15 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Impairment; Sleep Quality
MeSH Terms: conditions — Cognitive Dysfunction; Sleep Initiation and Maintenance Disorders | interventions — nicotinamide-beta-riboside; Niacinamide

STUDY DESIGN:
Intervention Model Description: A clinical trial, randomized controlled trial, double-blinded. Participants will be assigned to intervention (NR supplementation) or placebo groups.
Who Masked: Participant
Masking Description: Study participants and investigators will be blinded to group assignment. A statistician will assign participants into groups and a pharmacist will distribute treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention group will receive 500mg of NR twice daily
  Interventions: Dietary Supplement: Nicotinamide riboside
- Placebo (Placebo Comparator): Participants in the intervention group will receive 500mg of sham placebo twice daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide riboside — Nicotinamide riboside (NR) is a form of vitamin B3, which is found in fruits, vegetables, meat, and milk. NR is converted into nicotinamide adenosine dinucleotide NAD+. Low NAD+ levels have been linked to Alzheimer's disease and sleep disturbances.
  Other Names: NR, vitamin B3
  Arms: Intervention
Dietary Supplement: Placebo — The placebo pill will contain micro cellulose powder.
  Other Names: Placebo pill
  Arms: Placebo

SUMMARY:
Poor sleep quality and short sleep duration may be a mechanistic component of cognitive impairment in older adults, associated with a decline in brain-derived neurotrophic factor. Increasing the availability of nicotinamide adenine dinucleotide (NAD+) with supplementation of its precursor, nicotinamide riboside (NR), a form of vitamin B3 may increase the expression of brain-derived neurotrophic factor. This study proposes to examine the benefits of NR supplementation on sleep and cognitive function in older adults with comprehensive subjective and objective measures and to explore its impacts on serum brain-derived neurotrophic factor.

DETAILED DESCRIPTION:
Ten percent of adults aged ≥ 65 years and fifty percent of adults ≥ 85 years exhibit cognitive impairment. Dementia treatment cost $277 billion in 2018 and is predicted to surpass $500 billion with the aged population reaching 70 million by 2030 in America. In addition, 50% of older adults experience poor sleep quality, including fragmented nighttime sleep, reduced sleep efficiency, and earlier bedtime and wake-up times. Consequently, millions of Americans are at risk for both cognitive impairment, including Alzheimer's Disease and other dementias, and disrupted sleep. Sleep disruptions alter underlying circadian rhythms and synaptic plasticity in the hippocampus, as well as reduce expression of brain-derived neurotrophic factor (BDNF) - elements associated with impaired memory, dementia, and Alzheimer's Disease. Importantly, sleep disturbances and mild cognitive impairment may appear several years before the development of clinical dementia. Therefore, interventions that improve sleep may prevent cognitive impairment and would have substantial clinical importance. Pre-clinical animal models suggest that enhancing the availability of nicotinamide adenine dinucleotide (NAD+) may reduce cognitive decline and support sleep quality by boosting mitochondrial function and BDNF expression. Additionally, supplementation with NAD+ precursor nicotinamide riboside (NR), a form of vitamin B3, improves cognition in aged mice. The hypothesis for this study is that NR supplementation will enhance cognition by improving objective sleep duration and sleep quality in older persons. To test the hypothesis, this study will measure the benefits of NR supplementation on sleep and cognition in older Veterans and determine the role of BNDF as a potential biomarker of sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Sleep Quality. Pittsburgh Sleep Quality Index (PSQI) global score >5

Exclusion Criteria:

* Dementia. Veteran Affairs - St. Louis University Mental Status questionnaire (VA-SLUMS) score <20

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality Assessment | Change from baseline to endpoint at 12 weeks
  Sleep quality will be assessed with the Pittsburgh Sleep Quality Index , where global score >5 indicates poor sleep quality and global score <5 indicates good sleep quality.

SECONDARY OUTCOMES:
Cognitive function | Change from baseline to endpoint at 12 weeks
  Cognitive function will be assessed with the Veterans Affairs St. Louis University Mental Health Status (VA-SLUMS), which contains 11 items designed to measure orientation, memory, attention, and executive function. Scores range from 0-30 with categories of unimpaired, mildly impaired, and impaired.

OTHER OUTCOMES:
Biomarkers | Change from baseline to endpoint at 12 weeks
  Assessment of serum levels of BDNF, NfL, Aβ42/Aβ40 ratio, and p-tau as potential markers of cognition and sleep

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - State University of New York at Buffalo, Buffalo, New York
  - University at Buffalo State University of New York, Buffalo, New York
  - Buffalo Veteran Affairs Medical Center, Buffalo, New York

IPD SHARING:
Plan to Share IPD: Yes
All clinical information obtained from the participants will be contained in a password-protected secure database that has been designed specifically for the current research proposal. Published or reported results from this trial will not contain any personal information that could be linked to individuals. The data will be monitored routinely to maintain safety and productivity, as well as to assist with research dissemination annually.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Published or reported results from this trial will not contain any personal information that could be linked to individuals. De-identified data will be utilized for the publication of research findings in conferences, and scientific journals and will become available at the anticipated study completion (January 2025)
Access Criteria: All information from data collection forms and clinical databases will be linked with the study identification number, and only deidentified data will be released and analyzed. All research files and consent forms will be stored in locked cabinets and rooms and will only be accessible to research personnel. All data files related to this project are located on a secure server with password-protected access.